CLINICAL TRIAL: NCT03465644
Title: Comparison of Tailored Antiplatelet Therapy With Early Escalation and Late De-Escalation Strategy Versus Standard Dual Antiplatelet Therapy in Patients Undergoing Complex High-Risk Percutaneous Coronary Intervention
Brief Title: TAILored Versus COnventional AntithRombotic StratEgy IntenDed for Complex HIgh-Risk PCI
Acronym: TAILORED-CHIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duk-Woo Park, MD (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Duk-Woo Park, MD, Professor, Division of Cardiology, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2018-03
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Coronary Stenoses
Keywords: antithrombotic strategy; dual antiplatelet therapy
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored arm (Experimental): early (<6-month post-PCI) intensified (low-dose ticagrelor [120 mg loading, then 60 mg bid maintenance] and aspirin) and late (>6-month post-PCI) deescalated (clopidogrel alone) strategy
  Interventions: Drug: Tailored antithrombotic strategy
- Conventional arm (Active Comparator): clopidogrel + aspirin for 12months
  Interventions: Drug: Conventional antithrombotic strategy

INTERVENTIONS:
Drug: Tailored antithrombotic strategy — Low-dose (60mg) ticagrelor + aspirin for 6months and then clopidogrel alone for 6months
  Arms: Tailored arm
Drug: Conventional antithrombotic strategy — Clopidogrel + aspirin for 12months
  Arms: Conventional arm

SUMMARY:
This study evaluates the efficacy and safety of tailored antithrombotic therapy with early (<6-month post-PCI) intensified (low-dose ticagrelor [120 mg loading, then 60 mg bid maintenance] and aspirin) and late (>6-month post-PCI) deescalated (clopidogrel alone) strategy in patients undergoing high-risk complex PCI as compared with standard Dual Antiplatelet Therapy(aspirin and clopidogrel for 12 months).

ELIGIBILITY:
Inclusion Criteria:

1. Age 19 and more
2. Subjects who scheduled for percutaneous coronary intervention(PCI) with contemporary drug-eluting stent
3. Patients must have at least one of any features of complex high-risk anatomic, procedural, or clinical-related factors;

   * Clinical factors: diabetes, chronic kidney disease (i.e. creatinine clearance <60 mL/min), or low left ventricular ejection fraction (<40%) or
   * Lesion- or procedure-related factors: left main PCI, chronic total occlusion, bifurcation lesion requiring two-stent technique, severe calcification, diffuse long lesion (lesion length ≥ at least 30 mm), multi-vessel PCI (≥ 2 vessels requiring stent implantation), ≥3 requiring stent implantation, ≥ 3 lesions will be treated, or predicted total stent length for revascularization > 60 mm
4. The patient or guardian agreed to the study protocol and the schedule of clinical follow-up and provided informed, written consent, as approved by the appropriate institutional review board/ethical committee of the respective clinical site.

Exclusion Criteria:

1. Enzyme-positive Acute myocardial infarction (non-ST-elevation myocardial infarction (NSTEMI) or ST Elevation Myocardial Infarction (STEMI))
2. Contraindication to aspirin or P2Y12 inhibitors (ticagrelor or clopidogrel)
3. Use of Gp IIb/IIIa inhibitors at randomization
4. Cardiogenic shock
5. Treatment with only bare-metal stent (BMS) or balloon angioplasty during the index procedure.
6. Requirements for chronic oral anticoagulation (warfarin or Non-vitamin K antagonist oral anticoagulant (NOACs))
7. Active bleeding or extreme-risk for major bleeding (e.g. active peptic ulcer disease, gastrointestinal pathology with a high risk for bleeding, malignancies with a high risk for bleeding)
8. History of intracranial hemorrhage or intracranial aneurysm
9. Planned surgery within 180 days
10. Severe liver disease (ascites and/or coagulopathy) or Dialysis-dependent renal failure at screening
11. Platelet count <80,000 cells/mm3 or hemoglobin level <10 g/dL
12. At risk of bradycardia (subjects with sinus node dysfunction or atrioventricular block more than 2nd degree but without a permanent pacemaker)
13. Use of strong cytochrome P-450 3A inhibitor or inducers within 2 week of the date of enrollment

    : ketoconazole, clarithromycin, nefazodone, ritonavir, atazanavir, rifampin/rifampicin, rifabutin, dexamethasone, phenytoin, carbamazepine, phenobarbital
14. Pregnant and/or lactating women.
15. Concurrent medical condition with a life expectancy of less than 1 years
16. Active participation in another investigational study of a drug or device that has not completed the primary endpoint or follow-up period
17. Inability to provide written informed consent or participate in long-term follow-up

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2018 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Net clinical outcome | 1 year
  a net clinical outcome of all-cause death, myocardial infarction, stroke, stent thrombosis, urgent revascularization or clinically relevant bleeding [Bleeding Academic Research Consortium (BARC) 2, 3, or 5] at 12 months after randomisation

SECONDARY OUTCOMES:
Death | 1 year
  Efficacy outcomes: any, cardiovascular, or non-cardiovascular cause death
Myocardial infarction | 1 year
  Efficacy outcomes: any, periprocedural, or spontaneous Myocardial infarction
Stroke | 1 year
  Efficacy outcomes: any, ischemic, or hemorrhagic Stroke
Stent thrombosis | 1 year
  Efficacy outcomes
The rate of unplanned urgent repeat revascularization | 1 year
  Efficacy outcomes: any, target-vessel, or non-target-vessel Repeat revascularisation
Composite of ischemic clinical endpoints (all-cause death, myocardial infarction, stroke, stent thrombosis, or urgent revascularization) | 1 year
  Efficacy outcomes
Composite of hard clinical endpoints (all-caused death, myocardial infarction, or stroke) | 1 year
  Efficacy outcomes
BARC major bleeding (type 3 or 5 bleeding) | 1 year
  Safety outcomes: Bleeding Academic Research Consortium
TIMI major or minor bleeding | 1 year
  Safety outcomes: Thrombolysis In Myocardial Infarction
GUSTO moderate or severe bleeding | 1 year
  Safety outcomes: Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Coronary Arteries
ISTH major bleeding | 1 year
  Safety outcomes: International Society of Thrombosis and Hemostasis; PCI, percutaneous coronary intervention
Any major or minor bleeding | 1 year
  Safety outcomes

CONTACTS AND LOCATIONS:
Locations (22):
- South Korea (22):
  - Hallym University Sacred Heart Hospital, Anyang
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Gyeongsang National University Changwon Hospital, Changwon
  - Chungbuk National University Hospital, Cheonju
  - Gangwon National Univ. Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - Dong-A Medical Center, Pusan
  - Inje University Pusan Paik Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Bundang CHA Hospital, Seongnam
  - Seoul university Bundang hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic Univ. of Korea Eunpyeong St. Mary's hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - St.Carollo Hospital, Suncheon
  - The Catholic University of Korea, ST. Mary's Hospital, Suwon
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang DY, Wee SB, Ahn JM, Park H, Yun SC, Park KH, Kang SH, Suh J, Bae JW, Park S, Cho JH, Suh JW, Lee BK, Rha SW, Won H, Jang JS, Cho YR, Lee CH, Ahn YK, Oh JH, Bae JS, Park CS, Lee JB, Choi J, Lee SW, Her SH, Kwon O, Park SJ, Park DW. Temporal modulation of antiplatelet therapy in high-risk patients undergoing complex percutaneous coronary intervention: the TAILORED-CHIP randomized clinical trial. Eur Heart J. 2025 Aug 31:ehaf652. doi: 10.1093/eurheartj/ehaf652. Online ahead of print. PMID 40886179
- [Derived] Park H, Kang DY, Ahn JM, Yun SC, Park KH, Kang SH, Suh J, Bae JW, Park S, Cho JH, Suh JW, Lee BK, Rha SW, Won H, Jang JS, Kim MH, Lee CH, Ahn YK, Oh JH, Bae JS, Park CS, Choi J, Lee JB, Lee SW, Hur SH, Kwon O, Park SJ, Park DW, Tailored-Chip Trial Investigators OBOT. Temporal modulation (early escalation and late de-escalation) of antiplatelet therapy in patients undergoing complex high-risk PCI: rationale and design of the TAILORED-CHIP trial. EuroIntervention. 2024 Nov 4;20(21):e1355-e1362. doi: 10.4244/EIJ-D-24-00437. PMID 39492701